CLINICAL TRIAL: NCT00398853
Title: Chromium and Insulin Action
Brief Title: Effect of Chromium Picolinate on Insulin Sensitivity in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, William Cefalu, MD, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01DK060126 (NIH)
Record Dates: First submitted 2006-11-09; First posted 2006-11-14 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes
Keywords: insulin; glucose; chromium
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — picolinic acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chromium Picolinate (Experimental): Chromium
  Interventions: Dietary Supplement: chromium picolinate 1000 mcg daily vs placebo
- Placebo (Other): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: chromium picolinate 1000 mcg daily vs placebo — chromium picolinate 1000 mcg daily vs placebo
  Arms: Chromium Picolinate
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The effect of Chromium to improve glucose levels in diabetes is controversial. The hypothesis of the study was to evaluate the effect of supplementing the diet of individuals with Type 2 diabetes with chromium picolinate and assessing the effect of the supplementation on insulin sensitivity as assessed with hyperinsulinemic clamps

DETAILED DESCRIPTION:
Detailed Description:

The primary clinical strategy to improve metabolic control in patients with Type 2 diabetes consists of lifestyle modification combined with pharmacologic intervention. However, alternative strategies, e.g. nutritional supplementation with over-the-counter agents, are extensively practiced by a large number of patients and are frequently undertaken without first informing the medical provider. Unfortunately, considerable controversy exists regarding use of dietary supplements in subjects with diabetes because efficacy data for many of the supplements consists of only uncontrolled studies and anecdotal reports. As such, there is a paucity of data in humans in regard to the effect of most commercially available supplements to improve metabolic abnormalities.

One supplement that has attracted considerable clinical interest is chromium (Cr). However, routine use of Cr in subjects with diabetes is not currently recommended. In part, the controversy surrounding Cr supplementation stems from the lack of definitive randomized trials, the lack of "gold standard" techniques to assess glucose metabolism in the studies reported, the use of differing doses and formulation , and the study of heterogeneous study populations. As such, conflicting data has been reported that has contributed greatly to the confusion among healthcare providers concerning Cr supplementation. In order to provide a comprehensive clinical evaluation of Cr, we conducted a randomized, double-blinded, placebo-controlled trial in subjects with Type 2 diabetes. Individuals had baseline measures consisting of oral glucose tolerance testing, body fat and adiposity assessed, and then used established techniques to assess insulin sensitivity with hyperinsulinemic-euglycemic clamps. Individuals were evaluated for 6 months at which time repeat testing was done.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* On no meds to alter glucose metabolism
* age greater than 25 years old
* Fasting glucose greater than 125 mg/dl at screening

Exclusion Criteria:

* Subjects on insulin
* Sujbects on meds that alter glucose metabolism
* Use of glitazones
* C0-existing disorders in major organ systems such as heart, kidneys, liver

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-10; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity as assessed with hyperinsulinemic-euglycemic clamps | at study enpoints

SECONDARY OUTCOMES:
glucose control | at study endpoints
body weight and fat distribution, myocellular and intrahepatic lipid content as assessed with MRS scans | at study endpoints

CONTACTS AND LOCATIONS:
Overall Officials: William Cefalu, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Broskey NT, Obanda DN, Burton JH, Cefalu WT, Ravussin E. Skeletal muscle ceramides and daily fat oxidation in obesity and diabetes. Metabolism. 2018 May;82:118-123. doi: 10.1016/j.metabol.2017.12.012. Epub 2018 Jan 4. PMID 29307520
- [Derived] Cefalu WT, Rood J, Pinsonat P, Qin J, Sereda O, Levitan L, Anderson RA, Zhang XH, Martin JM, Martin CK, Wang ZQ, Newcomer B. Characterization of the metabolic and physiologic response to chromium supplementation in subjects with type 2 diabetes mellitus. Metabolism. 2010 May;59(5):755-62. doi: 10.1016/j.metabol.2009.09.023. Epub 2009 Dec 22. PMID 20022616